CLINICAL TRIAL: NCT06555068
Title: An Open-Label, Multi-Center Phase Ib/II Clinical Study Evaluating the Safety, Tolerability, Pharmacokinetics, and Preliminary Efficacy of HRS-6209 in Combination With Fulvestrant, Letrozole, HRS-8080, or HRS-1358 in Patients With Advanced Unresectable or Metastatic Breast Cancer
Brief Title: A Trial of HRS-6209 in Combination With Fulvestrant, Letrozole, HRS-8080, or HRS-1358 in Breast Cancer Patients
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Jiangsu HengRui Medicine Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HRS-6209-201
Record Dates: First submitted 2024-08-01; First posted 2024-08-15 (Actual); Last update posted 2025-06-22 (Actual); Status verified 2024-08

CONDITIONS: Advanced Unresectable or Metastatic Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Fulvestrant; Letrozole

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- Treatment group A: HRS-6209 in Combination with Fulvestrant (Experimental)
  Interventions: Drug: HRS-6209 in Combination with Fulvestrant
- Treatment group E: HRS-6209 in Combination with HRS-1358 (Experimental)
  Interventions: Drug: HRS-6209 in Combination with HRS-1358
- Treatment group B：HRS-6209 in Combination with Letrozole (Experimental)
  Interventions: Drug: HRS-6209 in Combination with Letrozole
- Treatment group C：HRS-6209 in Combination with HRS-8080 (Experimental)
  Interventions: Drug: HRS-6209 in Combination with HRS-8080
- Treatment group D：HRS-6209 in Combination with HRS-1358 (Experimental)
  Interventions: Drug: HRS-6209 in Combination with HRS-1358

INTERVENTIONS:
Drug: HRS-6209 in Combination with Fulvestrant — HRS-6209 in Combination with Fulvestrant
  Arms: Treatment group A: HRS-6209 in Combination with Fulvestrant
Drug: HRS-6209 in Combination with HRS-1358 — HRS-6209 in Combination with HRS-1358
  Arms: Treatment group E: HRS-6209 in Combination with HRS-1358
Drug: HRS-6209 in Combination with Letrozole — HRS-6209 in Combination with Letrozole
  Arms: Treatment group B：HRS-6209 in Combination with Letrozole
Drug: HRS-6209 in Combination with HRS-8080 — HRS-6209 in Combination with HRS-8080
  Arms: Treatment group C：HRS-6209 in Combination with HRS-8080
Drug: HRS-6209 in Combination with HRS-1358 — HRS-6209 in Combination with HRS-1358
  Arms: Treatment group D：HRS-6209 in Combination with HRS-1358

SUMMARY:
The study is being conducted to evaluate the safety, PK and efficacy of HRS-6209 in Combination with Fulvestrant, Letrozole, HRS-8080, or HRS-1358 for advanced unresectable or metastatic breast cancer

ELIGIBILITY:
Inclusion Criteria:

1. Females aged 18-75 years (inclusive);
2. ECOG performance status (PS) score of 0-1;
3. Patients with histopathologically confirmed metastatic or unresectable locally advanced breast cancer, histopathologically confirmed ER-positive or PR-positive;
4. Menopausal status:

   1. Having had bilateral oophorectomy, or aged ≥ 60 years old; or
   2. Aged < 60, natural menopause with E2 and FSH at postmenopausal levels; or
   3. Premenopausal or perimenopausal patients, but they should receive LHRH agonists during the study and the treatment should be initiated prior to study treatment.
5. Disease progression evidenced by imaging during or after the last systemic anti-tumor treatment prior to the first dose (limited to the efficacy expansion stage);
6. With at least one extracranial measurable target lesion at baseline per RECIST v1.1;
7. Life expectancy of > 3 months;
8. The functional level of organs must meet the following requirements :

   Absolute neutrophil count ≥ 1.5 × 109/L; Platelet count ≥ 90 × 109/L; Hemoglobin ≥ 10 g/dL; Normal blood creatinine or creatinine clearance ≥ 50 mL/min (calculated by standard Cockcroft-Gault formula); Serum albumin ≥ 3.0 g/dL; Total bilirubin ≤ 1.5 × upper limit of normal (ULN); Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤ 2.5 × ULN, or ≤ 5.0 × ULN for patients with liver metastasis; Prothrombin time (PT) and partial thromboplastin time (APTT) ≤ 1.5 × ULN; Urine protein < 2+ or 24-h urine protein < 1 g; Left ventricular ejection fraction (LVEF) ≥ 50%; QTcF ≤ 470 msec.
9. Female subjects of childbearing potential should agree to adopt effective contraceptive measures during the study period and within 6 months after the end of the study treatment; female subjects of childbearing potential must have a negative serum HCG test result within 7 days before enrollment in the study and must not be in the lactation;
10. Voluntarily participate in this clinical study, be willing and able to comply with procedures related to clinical visits and study, and understand and have signed written informed consent.

Exclusion Criteria:

1. With symptomatic visceral metastases deemed unfit for endocrine therapy by the investigator;
2. With active brain metastases, carcinomatous meningitis, spinal cord compression, or a history of primary tumors of the central nervous system;
3. History of clinically significant cardiovascular disease;
4. Abnormal ECG findings, which are judged by the investigator to be clinically significantand and need to intervene ;
5. With factors that affect oral medication, active gastrointestinal diseases, or other diseases that may obviously affect drug absorption, distribution, metabolism, or excretion;
6. With clinically significant endometrial abnormalities, including but not limited to endometrial hyperplasia and dysfunctional uterine bleeding;
7. Active infection or unexplained fever > 38.5 °C during the screening period or on the day of first dose;
8. With uncontrollable chronic systemic complications as judged by the investigator.
9. With active autoimmune diseases, history of immunodeficiency and history of autoimmune diseases, history of diseases or syndromes that require systemic corticosteroids or immunosuppressive drugs, other acquired (HIV infection) or congenital immunodeficiency, or history of organ transplantation (including allogeneic bone marrow transplantation);
10. With acute infection or active tuberculosis requiring medication.
11. With a known history of clinically significant liver disease, untreated active hepatitis;
12. Had other concurrent malignant tumors in the past 5 years;
13. Use of moderate and strong CYP3A4 inhibitors within 1 week or moderate and strong CYP3A4 inducers within 2 weeks prior to the first dose;
14. Use of any drugs with the risk of prolonging QT/QTc interval or causing torsade de pointes (TdP) within 4 weeks prior to the first dose, and with previous congenital QT interval prolongation syndrome or a family history of QT interval prolongation;
15. Pregnant or lactating women, or females planning to become pregnant during the study period;
16. With clear history of neural or mental disorders or with history of psychotropic abuse or drug abuse;

19) Subjects who are expected to receive other anti-tumor therapies or drugs during this study.

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 528 (Estimated)
Dates: Start 2024-08-12 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2026-08 (Estimated)

PRIMARY OUTCOMES:
DLT (dose-limiting toxicity)-Stage I (dose exploration) | 28 days after the first dose
MTD (maximum tolerated dose) -Stage I (dose exploration) | 28 days after the first dose
RP2D (recommended phase II dose) -Stage I (dose exploration) | 28 days after the first dose
(Serious) AEs-Stage I (dose exploration) | every week in Cycle 1 (28 days after the first dose), every 2 weeks in Cycle 2 (28 days after the second dose), every 4 weeks from Cycle 3 and thereafter (28 days after each dose), lasting about one year
ORR ( objective response rate )-Stage II (efficacy expansion) | every 8 weeks lasting about one year

SECONDARY OUTCOMES:
Cmax, ss (Stage I) | Cycle 1 (each cycle is 28 days) day 15、Cycle 2 (each cycle is 28 days) and Cycle 3 (each cycle is 28 days)
Tmax, ss (Stage I) | Cycle 1 (each cycle is 28 days) day 15、Cycle 2 (each cycle is 28 days) and Cycle 3 (each cycle is 28 days)
Cmin, ss(Stage I) | Cycle 1 (each cycle is 28 days) day 15、Cycle 2 (each cycle is 28 days) and Cycle 3 (each cycle is 28 days)
AUCss (Stage I) | Cycle 1 (each cycle is 28 days) day 15、Cycle 2 (each cycle is 28 days) and Cycle 3 (each cycle is 28 days)
ORR (objective response rate) (Stage I) | every 8 weeks lasting about one year
BOR (best overall response) (Stage I) | every 8 weeks lasting about one year
DoR (duration of response) (Stage I) | every 8 weeks lasting about one year
CBR (clinical benefit rate) (Stage I) | every 8 weeks lasting about one year
PFS (progression-free survival) (Stage I) | every 8 weeks lasting about one year
(Serious) AEs (Stage II) | every week in Cycle 1 (28 days after the first dose), every 2 weeks in Cycle 2 (28 days after the second dose), every 4 weeks from Cycle 3 and thereafter (28 days after each dose), lasting about one year
Cmax, ss (Stage II) | Cycle 1 (each cycle is 28 days) day 15、Cycle 2 (each cycle is 28 days) and Cycle 3 (each cycle is 28 days)
Tmax, ss (Stage II) | Cycle 1 (each cycle is 28 days) day 15、Cycle 2 (each cycle is 28 days) and Cycle 3 (each cycle is 28 days)
Cmin, ss(Stage II) | Cycle 1 (each cycle is 28 days) day 15、Cycle 2 (each cycle is 28 days) and Cycle 3 (each cycle is 28 days)
AUCss (Stage II) | Cycle 1 (each cycle is 28 days) day 15、Cycle 2 (each cycle is 28 days) and Cycle 3 (each cycle is 28 days)
BOR (best overall response) (Stage II) | every 8 weeks lasting about one year
DoR (duration of response) (Stage II) | every 8 weeks lasting about one year
CBR (clinical benefit rate) (Stage II) | every 8 weeks lasting about one year
PFS (progression-free survival) (Stage II) | every 8 weeks lasting about one year

CONTACTS AND LOCATIONS:
Locations (1):
- Fudan University Shanghai Cancer Center, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided